CLINICAL TRIAL: NCT01211678
Title: Biomarkers of Anti-TNF-α Therapy Efficacy in Rheumatoid Arthritis to Define Unresponsive Patients (BATTER-UP)
Brief Title: Biomarkers of Anti-TNF-α Therapy Efficacy in Rheumatoid Arthritis to Define Unresponsive Patients
Acronym: BATTER-UP
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Collaborators: Crescendo Biosciences (Unknown)
Responsible Party: Sponsor
Other Study IDs: 999RA002
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma.
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study was to validate the ability of an 8-gene biomarker set to differentiate between participants who met or did not meet European League Against Rheumatism (EULAR) Disease Activity Score (DAS)-28 Good Response criteria after treatment with anti-Tumor Necrosis Factor (TNF) therapy for 14 weeks in approximately 200 anti-TNF-naïve participants. The secondary objectives of this study was (i) to compare the behavior of the 8-gene marker set in participants who were anti-TNF naïve versus those who began their second anti-TNF treatment , (ii) to develop, maintain, and utilize a biorepository of serum, plasma, RNA, and deoxyribonucleic acid (DNA) samples for additional experiments and analyses and (iii) to discover novel genetic (DNA) predictors of response to anti-TNF therapy.

ELIGIBILITY:
Key Inclusion Criteria

To be eligible to participate in this study, candidates must meet the following eligibility criteria at the time of enrollment:

* Are willing and able to provide informed consent..
* Meet the ACR criteria for RA as determined by a rheumatologist who is board certified in Rheumatology or a member of the ACR.
* Have 4 or more tender and 4 or more swollen joints out of 28 joints as assessed by their treating rheumatologist or a trained joint assessor.
* Subjects are not taking any of the following treatments and/or have washed out for the minimum duration as defined below. If subjects are currently taking these treatments, must have been on a stable dosing regimen for the minimum duration as defined below:

  * Oral DMARDs (MTX, hydroxychloroquine, sulfasalazine, leflunomide, cyclosporine, azathioprine): on drug for at least 3 months and washed out or stable for at least 6 weeks prior to baseline sample collection.
  * Oral corticosteroids: washed out or stable AND ≤10 mg/day of prednisone equivalent for at least 4 weeks prior to baseline sample collection.
  * Intraarticular or parenteral corticosteroids: Washed out or stable for at least 4 weeks prior to baseline sample collection.
  * NSAIDs: Washed out or stable for at least 2 weeks prior to baseline sample collection.
* Are about to start treatment with an anti-TNF agent approved for the treatment of RA for the first time OR Have not, in the opinion of the treating rheumatologist, achieved or maintained an adequate response to treatment with their first anti-TNF agent (any anti-TNF agent approved for the treatment of RA), and have been prescribed a different anti TNF agent. Subjects who switch for any reason other than lack of efficacy will be excluded.

Key Exclusion Criteria

Candidates will be excluded from study entry if any of the following exclusion criteria exist at the time of enrollment:

* Any medical condition that would preclude safe use of an anti-TNF agent for at least 14 weeks.
* Previous participation in the present study as a subject in the anti-TNF-naïve group.
* Prior exposure to 2 or more anti-TNF agents.
* Prior exposure to Orencia (abatacept, or CTLA4-Ig) and/or Rituxan (anti CD20), or other biologic therapy for RA or other diseases.

Note: Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who meet American College of Rheumatology (ACR) criteria for rheumatoid arthritis (RA) and who, in the opinion of their treating rheumatologist, are not adequately treated with existing therapy and should begin treatment with either an anti TNF agent for the first time or with a different anti-TNF agent.
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2010-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Validation of the ability of an 8-gene biomarker set to differentiate between participants who meet or do not meet EULAR DAS-28 Good response criteria after treatment with anti-TNF therapy | 14 weeks

SECONDARY OUTCOMES:
Comparison of the behavior of the 8-gene marker set in participants who are anti-TNF naïve versus those who begin their second anti-TNF treatment | 14 weeks
Development, maintenance, and utilization of a biorepository of serum, plasma, RNA, and deoxyribonucleic acid (DNA) samples for additional experiments and analyses. | 14 weeks
Discovery of novel genetic (DNA) predictors of response to anti-TNF therapy. | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (30):
- United States (30):
  - Research Site, Murrieta, California
  - Research Site, Longmont, Colorado
  - Research Site, Lewes, Delaware
  - Research Site, Dunedin, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orange Park, Florida
  - Research Site, Morton Grove, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Plymouth, Massachusetts
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Berkeley Heights, New Jersey
  - Research Site, Summit, New Jersey
  - Research Site, Floral Park, New York
  - Research Site, Orchard Park, New York
  - Research Site, Smithtown, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Mayfield Village, Ohio
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Edmund, Oklahoma
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Mrytle Beach, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, San Anotnio, Texas
  - Research Site, Burke, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
  - Research Site, Franklin, Wisconsin